CLINICAL TRIAL: NCT01635283
Title: A Phase II Clinical Trial Evaluating Autologous Dendritic Cells Pulsed With Tumor Lysate Antigen for the Treatment of Low-grade Glioma
Brief Title: Vaccine for Patients With Newly Diagnosed or Recurrent Low-Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-002665; NCI-2012-00980 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-06-22; First posted 2012-07-09 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2016-05

CONDITIONS: Adult Diffuse Astrocytoma; Adult Mixed Glioma; Adult Oligodendroglioma; Recurrent Adult Brain Tumor; Adult Oligoastrocytoma
MeSH Terms: conditions — Astrocytoma; Glioma; Oligodendroglioma; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (tumor lysate-pulsed autologous dendritic cells) (Experimental): Patients receive autologous glioma tumor lysate-pulsed autologous dendritic cell vaccine ID on days 0, 14, and 28.
  Interventions: Biological: tumor lysate-pulsed autologous dendritic cell vaccine; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: tumor lysate-pulsed autologous dendritic cell vaccine — Given ID
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
The primary purpose of this phase II clinical trial is to determine the safety and effect on survival of patients autologous dendritic cells pulsed with autologous tumor lysate as a treatment for low-grade glioma patients. Other goals of this study are to determine if the vaccine can cause an immune response against patients' cancer cells and slow the growth of their brain tumors

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the 5-year progression-free survival (PFS), using intradermal injections of autologous dendritic cells harvested from peripheral blood precursors and pulsed (co-cultured) with tumor lysate derived from surgical tissues in patients with low-grade gliomas.

SECONDARY OBJECTIVES:

I. To monitor overall survival (OS), and cellular immune responses in brain tumor patients injected with tumor lysate-pulsed dendritic cells.

OUTLINE:

Patients receive tumor lysate-pulsed autologous dendritic cell vaccine intradermally (ID) on days 0, 14, and 28.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed or recurrent glioma of World Health Organization (WHO) grade II (astrocytoma, oligodendroglioma, and/or oligoastrocytoma) will be eligible for this protocol
* Patients must have had surgical resection at University of California, Los Angeles (UCLA), for which a separate informed consent was signed for the collection of their tumor prior to surgery
* After surgery, a pathological diagnosis of low-grade glioma (WHO grade II) will need to be established
* Patients must be able to read and understand the informed consent document; patients must sign the informed consent indicating that they are aware of the investigational nature of this study.
* Patients must have a Karnofsky performance status (KPS) rating of >= 60 prior to initiating treatment; patients may be enrolled at a KPS of < 60 if it is felt that the patient will have adequate opportunity to recover to a KPS of >= 60 by the initiation of treatment
* Hemoglobin >= 9 gm%
* Absolute granulocyte count >= 1,500
* Platelet count >= 100,000/microliter (uL)
* Serum glutamic pyruvate transaminase (SGPT), serum glutamic oxaloacetic transaminase (SGOT) =< 2.5 times institutional normals
* Bilirubin =< 1.5mg%
* Blood urea nitrogen (BUN) or creatinine =< 1.5 times institutional normals

Exclusion Criteria:

* Subjects with an active infection
* Inability to obtain informed consent because of psychiatric or complicating medical problems
* Unstable or severe intercurrent medical or psychiatric conditions as determined by the Investigator
* Females of child-bearing potential who are pregnant or lactating or who are not using approved contraception
* History of immunodeficiency (e.g., human immunodeficiency virus [HIV]) or autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, vasculitis, polymyositis-dermatomyositis, scleroderma, multiple sclerosis, or juvenile-onset insulin-dependent diabetes) that may be exacerbated by immunotherapy
* Subjects with organ allografts
* Inability or unwillingness to return for required visits and follow-up exams
* Subjects who have an uncontrolled systemic malignancy that is not in remission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-01-10 (Actual); Primary Completion 2016-05-13 (Actual); Study Completion 2016-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Prins, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: 1/2012 - 8/2015 Types of location: Medical clinic
Pre-assignment Details: Study enrollment patients must satisfy inclusion criteria, screening evaluations (vital signs, history, physical, neurological exams, Karnofsky Performance Scale, brain MRI , urinalysis, complete blood count, differential, platelets, coagulation tests), underwent leukapheresis, and had suitable Dendritic Cell (DC) Vaccine manufactured for them.
Period: Overall Study
Arm/Group | Treatment (Tumor Lysate-pulsed Autologous Dendritic Cells)
Started | 5
Completed | 1
Not Completed | 4
Not completed — Tumor Progression | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Tumor Lysate-pulsed Autologous Dendritic Cells)
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (21.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) of Low Grade Glioma Patients Treated With Autologous Dendritic Cells Pulsed With Autologous Tumor Lysate
Description: a Kaplan-Meier curve of the PFS of our trial patients was created and compared to the PFS of control patients matched for tumor grade, recurrence number, IDH1 status and 1p/19q status.
Time Frame: Each case was assessed from the baseline date of surgery to MRI evidence of tumor progression through study completion, up to 44 months.
Population: Completed the maximum time allowed on study without being affected by Tumor Recurrence or Progression.
Measure: Number; unit: participants
Arm/Group | Treatment (Tumor Lysate-pulsed Autologous Dendritic Cells)
Number analyzed (Participants) | 5
participants
  0-6 months | 0
  7-12 months | 1
  13-18 months | 1
  19-24 months | 1
  25-30 months | 0
  >30 months | 2

2. Secondary Outcome: Overall Survival (OS)
Description: From date of enrollment until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 100 months. a Kaplan-Meier curve of the OS of our trial patients was created and compared to the OS of control patients matched for tumor grade, recurrence number, IDH1 status and 1p/19q status.
Time Frame: The timeframe for OS was from the date of surgery until the date of death from any cause, up to 44 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tumor Lysate-pulsed Autologous Dendritic Cells)
Number analyzed (Participants) | 5
Participants
  Deceased | 0
  Alive | 5
  Lost to Follow-Up | 0
  Withdrawal by Subject | 0

3. Secondary Outcome: Anti-tumor Immune Responses
Description: Tumor and peripheral blood samples were collected from each of the participants and analyzed for the following biomarkers:
  IDH1-specific antibodies CD8, PD-1, and PD-L1 content, and correlations among those three biomarkers Mutation analysis/sequencing
Time Frame: Tumor for analysis (CD8, Programmed Death (PD)-1, PD-L1, mutation analysis) was collected at the vaccine-related surgery shortly after enrollment. Blood for analysis (IDH1-specific antibodies) was collected at Day 0, before the first vaccine injection.
Population: Quantitative multiplex immuno-histochemical (IHC) of pre-treatment glioma microenvironment of IDH1-specific antibodies
Measure: Mean (Standard Deviation); unit: percentage of cells per field
Arm/Group | %CD8+/Field | %PD-1+/Field | %PD-L1+/Field
Number analyzed (Participants) | 5 | 5 | 5
percentage of cells per field | 1.26 (1.03) | 1.35 (1.04) | 6.76 (3.30)

ADVERSE EVENTS:
Time Frame: The timeframe for adverse event reporting was from the day of the first vaccine treatment until the patient discontinued the study for any reason, up to 44 months.
Arm/Group | Treatment (Tumor Lysate-pulsed Autologous Dendritic Cells)
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tumor Lysate-pulsed Autologous Dendritic Cells) (N=5)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (2)
Dysphasia (Nervous system disorders) | 1 (1)
Visual Distortions (Nervous system disorders) | 1 (1)
cognitive slowness (Nervous system disorders) | 1 (1)
Fractures (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Squamous cell carcinomas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Upper respritory infection (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Headache (General disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Rhinorrhea (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes